CLINICAL TRIAL: NCT07071324
Title: CF Wellness Program: ORBIT Phase 2 Pilot RCT
Brief Title: CF Wellness Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Boston Children's Hospital, Boston, MA, USA (Other); National Jewish Health (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00496586
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis (CF); Fatigue; Sleep Quality; Insomnia
Keywords: Cystic Fibrosis (CF); Fatigue; Sleep Quality; Physical Activity; Insomnia; Cognitive Behavioral Therapy; Sedentary
MeSH Terms: conditions — Cystic Fibrosis; Fatigue; Sleep Initiation and Maintenance Disorders; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Adults With Cystic Fibrosis (AWCF) randomized to the intervention will receive the CFWP written materials and be offered up to 8 coaching sessions tailored to fatigue, physical activity, and mental well-being. The sessions will last approximately 45 - 60 minutes and be delivered either by web-based video chat (e.g., Zoom) or by telephone.
  Interventions: Behavioral: CF Wellness Program
- Usual Care (No Intervention): Usual clinical care

INTERVENTIONS:
Behavioral: CF Wellness Program — Intervention modules are 1) Introduction & Fatigue Explained, 2) Finding Balance between Activity & Rest, 3) Physical Activity, Self-Review & Planning, 4) Improving Your Sleep, 5) Managing Emotions, 6) Changing Less Helpful Thoughts, 7) Learning to Relax & Manage Stress, and 8) Accessing Social Support and Preparing for the Future.
  Arms: Treatment Group

SUMMARY:
This study is a pilot randomized control trial (RCT; N=80) comparing the Cystic Fibrosis Wellness Program (CFWP) to usual care (UC) to evaluate (1) Intervention Adherence (completion of the CFWP Coaching Sessions) (2) Study Retention (completion of the Week 15 assessment) and (3) Data Quality (valid daytime and nighttime fitness tracker data). A secondary aim is to gather preliminary data to determine if the CFWP has a clinically significant signal over usual care to improve fatigue, sleep, and physical activity (PA) and reduce sedentary behavior.

DETAILED DESCRIPTION:
Highly effective modulator therapy (HEMT) has improved lung health for many adults with cystic fibrosis (CF), but does not appear to have translated into improved fatigue, sleep, or physical activity (PA). A study of 236 adults with CF (86% of whom were taking HEMT) found that 43% experienced elevated fatigue, while 63% reported poor sleep quality. Fatigue, poor sleep, and less PA are associated with worse physical and mental health outcomes, such as respiratory symptoms, lung function, depression, and anxiety. Cognitive behavioral therapy (CBT) is a well-established treatment for insomnia, pain, and mood disorders, with emerging data that it helps with fatigue. Similarly, increasing PA reduces fatigue and improves sleep. There is no research evaluating whether CBT or PA improves fatigue or sleep for adults with CF. Investigators developed a CBT+PA intervention for adults with CF and fatigue, known as the CF Wellness Program (CFWP), which includes written materials and up to eight virtual sessions with a Coach. The goal of the proposed pilot study is twofold. First, to evaluate session attendance and determine if research-quality fitness tracker data can be collected to objectively measure sleep and PA. Second, investigators will gather preliminary data to determine if the CFWP has a clinically significant signal over usual care to improve fatigue, sleep, and PA and reduce sedentary behavior. This study will enroll 80 adults with CF and fatigue. After completing the baseline assessment, half the participants will be randomized to receive the CFWP and half will not. The follow-up assessment will be collected at Week 15.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Documentation of CF diagnosis in the medical record
3. Score of >4 on the Fatigue Severity Scale
4. Access to a smartphone, tablet, and/or computer with access to internet
5. Ability to understand/read/speak English
6. Receives CF care at a participating CF Center

Exclusion Criteria:

1. Pulmonary exacerbation (physician determined and may include oral antibiotics, IV antibiotics, hospitalization) ±14 days of enrollment
2. Pregnant or <6 months post-partum (self-reported)
3. Contraindication to light physical activity (as determined by the treating physician and may include pulmonary, cardiovascular, or musculoskeletal contraindications)
4. Participated in the CFWP Feasibility Study
5. Currently enrolled in another interventional trial
6. Unavailable to complete coaching sessions within the study timeframe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Intervention Adherence as assessed by the number of CFWP participants | Up to 15 weeks
  The number of participants randomized to receive the CFWP who complete all 8 coaching sessions.
Participant Retention as assessed by the number of participants completing the week 15 assessment survey | Week 15
  The number of participants across both study groups who complete the week 15 assessment survey.
Fitness Tracker Data Quality as assessed by the number of participants who have valid activity and sleep data. | Baseline, Week 15
  The number of participants who have valid sleep and activity data at the baseline and week 15 assessment. Valid physical and sleep activity was defined as >10 hours of collected data across 4 days, including 1 weekend day and overnight.

SECONDARY OUTCOMES:
Fatigue as assessed by the Functional Assessment of Chronic Illness-Fatigue (FACIT-F) | Baseline, Week 15
  The number of CFWP participants reporting clinically improved fatigue compared to UC participants at the week 15 assessment. The FACIT-F is a 14-question instrument used to assess self-reported fatigue. Scores range from 0-52, with a score of <34 indicating clinically significant fatigue. Lower scores indicate higher fatigue. Clinically improved fatigue is defined as a ≥4 points increase in the FACIT-F or no longer having fatigue (FACIT-F ≥34).
Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 15 weeks
  The PSQI is a 19-item questionnaire that measures an individual's quality of sleep over the last month. Scores range from 0 to 21, with a score >5 indicative of poor sleep quality.
Sleep Quality as assessed by the Insomnia Severity Index (ISI) | Baseline, 15 weeks
  The ISI is a 7-item scale measuring the impact of insomnia in the past month. Total score ranging from 0 to 28, scores are categorized to indicate the severity of insomnia, ranging from no clinically significant insomnia (0-7) to severe insomnia (22-28). Higher score more severe insomnia.
Sleep patterns as assessed by the Consensus Sleep Diary - Core (CSD-C). | Baseline, 15 weeks
  The CSD-C is a 9-item self-reported diary of sleep activity to determine patterns such as good sleeper or insomnia.
Participant physical activity levels assessed by fitness tracker data | Baseline, Week 15
  Sedentary behavior will be defined as averaging <5000 steps/day, physically active will be defined as averaging >7500 steps/day, and consistent physical activity will be defined as a greater reduction in the daily step count standard deviation at baseline compared to the week 15 assessment.
Physical activity (PA) as assessed the International Physical Activity Questionnaire (IPAQ) - Short Form. | Baseline, Week 15
  The IPAQ is a 7-item self-report on physical activity. Minutes represent the amount of energy expended carrying out physical activity. A higher score represents a better outcome. Scores can range from 0 to 10,080

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Riekert, PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes